CLINICAL TRIAL: NCT02107599
Title: A Study to Evaluate the Improvement in Reader Accuracy When Using a Read Method That Incorporates Commercially Available Quantitative Analysis Software as an Adjunct to the Clinical Visual Interpretation of Amyvid Brain Scans
Brief Title: The Feasibility of Florbetapir Quantitation in Europe
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-QP02
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Results first posted 2015-07-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-06

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — florbetapir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physician Readers (Experimental): Physician readers will interpret Amyvid scans using qualitative analysis followed by the use of quantitation. No subjects will be exposed to Florbetapir(18F) as part of this study.
  Interventions: Drug: Florbetapir (18F)

INTERVENTIONS:
Drug: Florbetapir (18F) — No Florbetapir (18F) will be administered in this study.
  Other Names: Florbetapir F 18; Amyvid; 18F-AV-45

SUMMARY:
This study will evaluate whether the addition of quantitation as an adjunct to visual interpretations significantly improves the accuracy of Amyvid scan interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Readers have undergone Amyvid reader training
* Readers have not more than minimal experience with quantitation of amyloid PET scans

Exclusion Criteria:

* Readers have previously been trained to quantitate amyloid PET scans

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals, Inc.
Locations (1):
- Research Site, Leiden, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- Florbetapir PET Scans: No subjects were enrolled in this study. Readers interpreted 96 Florbetapir scans from subjects enrolled in previous studies (A16[NCT01447719] and A17[NCT01400425]). Scans used in the study included 46 scans with autopsy (A16) and 50 randomly selected non-autopsy scans (A17).
Period: Overall Study
Arm/Group | Florbetapir PET Scans
Started | 96
Completed | 96
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Florbetapir PET Scans
Number analyzed (Participants) | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.9 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 92
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1
  Black or African American | 5
  White | 89
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 96

OUTCOME MEASURES:

1. Primary Outcome: Change in Reader Accuracy After Application of Quantitation Software
Description: Evaluate whether the use of quantitation software improves florbetapir (18F) scan interpretation by using the net reclassification index (NRI). The NRI is a prospective measure that quantifies the correctness of upward and downward reclassification or movement of predicted probabilities as a result of adding a new marker. NRI Values >0 indicate an improvement in scan interpretation accuracy and values <0 indicate a decline in scan interpretation accuracy after application of quantitation software.
  NRI = [P(up,event)-P(down,event)]-[P(up,nonevent)-P(down,nonevent)] Where P(up,event) = # events up/# events P(down,event) = # events down/# events P(up,nonevent) = # nonevents up/# nonevents P(down,nonevent) = # nonevents down/# nonevents and events: true positive case nonevents: true negative case up: scan change from negative to positive down: scan change from positive to negative
  Only the 46 scans with autopsy from A16 are used for this outcome measure.
Time Frame: Scan acquired 50-60 minutes post injection
Measure: Number; unit: Net Reclassification Index
Groups:
- Physician Readers: All 21 physician readers.
Arm/Group | Physician Readers
Number analyzed (Participants) | 46
Net Reclassification Index | 0.0746
Statistical Analysis 1: Comparison: Physician Readers; Test type: Superiority or Other; p = 0.0001, Asymptotic Z-test

2. Secondary Outcome: Change in Scan Interpretation Reliability After Application of Quantitation Software
Description: as for outcome 1
Time Frame: Scan acquired 50-60 minutes post injection
Measure: Number (95% Confidence Interval); unit: Fleiss Kappa
Groups:
- All Study Cases: All 96 scans from A16 and A17.
- Autopsy Cases: Only 46 autopsy scans from A16.
- Non-autopsy Cases: Only 50 non-autopsy scans from A17.
Arm/Group | All Study Cases | Autopsy Cases | Non-autopsy Cases
Number analyzed (Participants) | 96 | 46 | 50
Fleiss Kappa
  Kappa VisQ | 0.73 [0.712 to 0.740] | 0.72 [0.703 to 0.743] | 0.73 [0.709 to 0.747]
  Kappa Qualitative | 0.66 [0.647 to 0.675] | 0.66 [0.644 to 0.684] | 0.66 [0.638 to 0.676]
  Change in Kappa | 0.06 [0.017 to 0.112] | 0.06 [-0.015 to 0.132] | 0.07 [0.008 to 0.133]
Statistical Analysis 1: Comparison: All Study Cases; Evaluate whether the VisQ interpretation significantly improves the reliability of Amyvid Scan interpretation; Test type: Superiority or Other; p = 0.0060, Monte Carlo test
Statistical Analysis 2: Comparison: Autopsy Cases; Evaluate whether the VisQ interpretation significantly improves the reliability of Amyvid Scan interpretation; Test type: Superiority or Other; p = 0.1229, Monte Carlo test
Statistical Analysis 3: Comparison: Non-autopsy Cases; Evaluate whether the VisQ interpretation significantly improves the reliability of Amyvid Scan interpretation; Test type: Superiority or Other; p = 0.0260, Monte Carlo test

ADVERSE EVENTS:
Time Frame: No subjects received florbetapir in this study. This study consisted of re-reads of scans previously acquired in other clinical studies (A16, and A17).
Arm/Group | Florbetapir PET Scans
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes